CLINICAL TRIAL: NCT03663803
Title: Effectiveness of a Brief Theory-based Health Promotion Intervention Among Adults at High Risk of Type 2 Diabetes: One-year Results From a Randomised Trial in a Community Setting
Brief Title: Live Your Life Without Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-02-3065
Record Dates: First submitted 2018-08-29; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group received the offer of four 2h group sessions during five weeks, and two further sessions after one and six months. The attendance rates of the sessions were 95%, 88%, 87%, 73%, 67% and 51%, respectively. The course was delivered by health care staff in the Holstebro Health Care Centre, including a dietitian and an occupational therapist, both with health pedagogic competences. It was delivered to seven intervention groups, which varied in size from 5 to 15 participants.
  Interventions: Behavioral: Brief theory-based health promotion intervention (group-based)
- Control (No Intervention): Usual practice

INTERVENTIONS:
Behavioral: Brief theory-based health promotion intervention (group-based) — The intervention is depicted using a PaT Plot in the published paper: Juul, L et al. Effectiveness of a brief theory-based health promotion intervention among adults at high risk of type 2 diabetes: One-year results from a randomised trial in a community setting. Primary Care Diabetes 1 0 ( 2 0 1 6 ) 111-120.
  Arms: Intervention

SUMMARY:
Aim: To examine the effect of a brief theory-based health promotion intervention delivered in the community on health behaviour and diabetes-related risk factors among Danish adults at high risk of diabetes.

Methods: A randomised trial was conducted among 127 individuals aged 28 to 70 with fasting plasma glucose: 6.1-6.9 mmol/l and/or HbA1c : 6.0-<6.5% (42- < 48 mmol/mol) recruited from general practice in Holstebro, Denmark. Participants were randomised to a control group or to receive the intervention delivered over four 2 h group sessions during five weeks, and two further sessions after one and six months. Questionnaire data and clinical measures were collected at baseline, three months and one year after intervention.

ELIGIBILITY:
Inclusion Criteria:

* resident in the Municipality of Holstebro
* aged <70 years
* a measurement of fasting plasma glucose: 6.1-6.9 mmol/l (the thresholds for Impaired Fasting Glucose according to clinical guidelines) and/or HbA1c : 6.0-<6.5% (42- <48 mmol/mol) within the previous six months.

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-01-19 (Actual); Primary Completion 2013-01-09 (Actual); Study Completion 2013-01-09 (Actual)

PRIMARY OUTCOMES:
weight | baseline to one-year follow-up
  change in weight / the proportion with weight reduction >5% of baseline weight at one-year
total-fat intake <30% of energy intake | change from baseline to one-year follow-up
  Information on diet was obtained using a validated self-administrated 198-item food frequency questionnaire (FFQ), the Inter99 FFQ. Portion size was set according to gender. Daily nutrient intake was translated into energy intake and nutrient intake using the Danish Food Com- position Databank (version 7.01) and the software program FoodCalc version 1.3
saturated-fat intake <10% of energy intake | change from baseline to one-year follow-up
  Information on diet was obtained using a validated self-administrated 198-item food frequency questionnaire (FFQ), the Inter99 FFQ. Portion size was set according to gender. Daily nutrient intake was translated into energy intake and nutrient intake using the Danish Food Com- position Databank (version 7.01) and the software program FoodCalc version 1.3
fibre-intake ≥15g/1000kcal changes in physical activity level. | change from baseline to one-year follow-up
  Information on diet was obtained using a validated self-administrated 198-item food frequency questionnaire (FFQ), the Inter99 FFQ. Portion size was set according to gender. Daily nutrient intake was translated into energy intake and nutrient intake using the Danish Food Com- position Databank (version 7.01) and the software program FoodCalc version 1.3
changes in physical activity. | change from baseline to one-year follow-up
  Physical activity was measured using the International Physical Activity Questionnaire (IPAQ). Increased MET (min/week)=increased physical activity

SECONDARY OUTCOMES:
patient activation | change from baseline to one-year follow-up
  patient activation was measured using the Patient Activation Measure (PAM)
waist circumference | change from baseline to one-year follow-up
  Waist circumference was recorded as the average of two measurements of waist circumference using a tape measure halfway between the lowest point of the rib cage and the anterior supe- rior iliac crests when standing.
total energy intake | change from baseline to one-year follow-up
  Information on diet was obtained using a validated self-administrated 198-item food frequency questionnaire (FFQ), the Inter99 FFQ. Portion size was set according to gender. Daily nutrient intake was translated into energy intake and nutrient intake using the Danish Food Com- position Databank (version 7.01) and the software program FoodCalc version 1.3
blood pressure, systolic and diastolic | change from baseline to one-year follow-up
  Systolic and diastolic blood pressure was calculated as the mean of three measurements performed after at least 10 min rest, while participants were seated with the cuff on the right arm at the level of the heart.
HbA1c | change from baseline to one-year follow-up
  Blood tests were analysed in a central laboratory.
cholesterol | change from baseline to one-year follow-up
  Total, LDL, HDL, Blood tests were analysed in a central laboratory.